CLINICAL TRIAL: NCT01784965
Title: Addition of a Glucagon-like Peptide-1 to a Calorie Restricted Diet Augments Weight Loss and Decreases Risk of Type 2 Diabetes and Cardiovascular Disease.
Brief Title: Liraglutide and a Calorie Restricted Diet Augments Weight Loss and Decreases Risk of Type 2 Diabetes and CVD.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gerald M Reaven, Professor Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17394
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Pre-diabetes; Older Adults
MeSH Terms: conditions — Glucose Intolerance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Both groups receive dietary weight loss intervention In addition one group received liraglutide and one group received placebo
  Interventions: Drug: Placebo
- liraglutide (Active Comparator): Both groups receive dietary weight loss intervention In addition one group received liraglutide and one group received placebo
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Dosing begins at 0.6 mg subcutaneous injection and increases each week, to 1.2 mg and maximum dose of 1.8 mg.
  Other Names: Victoza
  Arms: liraglutide
Drug: Placebo — Double blinded will receive study pen with same dosing instructions starting at 0.6 mg, and each week increase to 1.2 mg and finally 1.8 mg at week three.
  Arms: placebo

SUMMARY:
The goal of this study is to evaluate the hypothesis that the addition of liraglutide, a long-acting glucagon-like peptide 1 (GLP-1) analogue, to a calorie-restricted diet will lead to greater weight loss than will a calorie-restricted diet alone in subjects who are older (50 to 60 years of age), overweight/obese, and prediabetic. These individuals have been selected for study because they are at greatly increased risk to develop type 2 diabetes (2DM) and cardiovascular disease (CVD), and it is hypothesized that the addition of liraglutide to a calorie-restricted diet will significantly decrease risk of these adverse outcomes.

There is considerable evidence that GLP-I compounds, including liraglutide, improve glycemic control in patients with manifest 2DM. However, there is relatively little information as to the potential utility of these compounds in nondiabetic individual at greatly increased risk of 2DM and CVD. This research proposal is aimed at providing some of this information by quantifying the effects of liraglutide, a long-acting GLP-1 analogue, on weight loss, insulin secretion, insulin action, and multiple CVD risk factors in a very high risk group-older, overweight/obese, prediabetic individuals. Furthermore, by using specific methods, not surrogate estimates, and avoiding the confounding effects of glucotoxicity, it will be possible to gain new insights into the effects of GLP-1 on insulin secretion and insulin action.

ELIGIBILITY:
Inclusion Criteria:

IFG, or IGT BMI 27.0-37.0 kg/m2

Exclusion Criteria:

DM, CAD, severe anemia, kidney or liver disease, hx of pancreatitis, gallstones, ETOH abuse, personnel or family history of medullary thyroid carcinoma or MEN-2

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald M Reaven, M.D., Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Liu A, Ariel D, Abbasi F, Lamendola C, Grove K, Tomasso V, Reaven G. Pancreatic beta cell function following liraglutide-augmented weight loss in individuals with prediabetes: analysis of a randomised, placebo-controlled study. Diabetologia. 2014 Mar;57(3):455-62. doi: 10.1007/s00125-013-3134-3. Epub 2013 Dec 11. PMID 24326527
- [Derived] Kim SH, Abbasi F, Lamendola C, Liu A, Ariel D, Schaaf P, Grove K, Tomasso V, Ochoa H, Liu YV, Chen YD, Reaven G. Benefits of liraglutide treatment in overweight and obese older individuals with prediabetes. Diabetes Care. 2013 Oct;36(10):3276-82. doi: 10.2337/dc13-0354. Epub 2013 Jul 8. PMID 23835684

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 person qualified and enrolled in study but dropped out before being randomized to either group. Therefore is not counted in placebo or liraglutide group.
Groups:
- Placebo: Both groups receive dietary weight loss intervention In addition one group received liraglutide and one group received placebo
  Placebo: Double blinded study. Participants will receive study pen with dosing instructions starting at 0.6 mg, and each week increase to 1.2 mg and finally 1.8 mg at week three.
- Liraglutide: Both groups receive dietary weight loss intervention In addition one group received liraglutide and one group received placebo
  Liraglutide: Double Blinded study. Participants will receive a study pen with dosing instructions: Dosing begins at 0.6 mg subcutaneous injection and increases each week, to 1.2 mg and maximum dose of 1.8 mg.
Period: Overall Study
Arm/Group | Placebo | Liraglutide
Started | 33 | 35
Completed | 27 | 24
Not Completed | 6 | 11
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Adverse Event | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Liraglutide | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8) | 58 (7) | 58 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (3.5) | 31.9 (2.7) | 31.9 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight Reported at 14 Weeks
Description: Change in weight with caloric restriction plus liraglutide vs. caloric restriction and placebo over 14 weeks.
Time Frame: Baseline and 14 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | Liraglutide
Number analyzed (Participants) | 27 | 24
kg | -3.3 [-4.1 to -2.5] | -6.8 [-7.8 to -5.9]
Statistical Analysis 1: Comparison: Placebo vs Liraglutide; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Glucose-stimulated Insulin Secretion in Insulin AUC, Pmol/1x 4H
Description: Absolute change in glucose-stimulated insulin secretion (GS-IS) associated with caloric restriction plus liraglutide vs. caloric restriction and placebo at 14 weeks
Time Frame: Baseline, 14 weeks
Measure: Mean (95% Confidence Interval); unit: pmol/l x4 h
Arm/Group | Placebo | Liraglutide
Number analyzed (Participants) | 27 | 24
pmol/l x4 h | -7.3 [-17 to 2] | 34 [21 to 48]

3. Secondary Outcome: Insulin Resistance in the Liraglutide vs.Placebo Group After Calorie Restriction
Description: Mean (+/- SD) change in insulin resistance associated with caloric restriction plus liraglutide vs. caloric restriction and placebo.
Time Frame: Baseline, 14 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Liraglutide
Number analyzed (Participants) | 27 | 24
mg/dL | 2.8 (35.9) | -57.5 (44.2)

ADVERSE EVENTS:
Groups:
- Liraglutide: Intolerable gastrointestinal side effects 3/35 injection site reaction 2/35 pneumonia 1/35 gallstone 1/35 fall 1/35
- Placebo: 0/33 0/33 0/33 0/33 0/33
Arm/Group | Liraglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 8/35 | 0/33
Other Adverse Events (participants affected / at risk) | 3/35 | 6/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=35) | Placebo (N=33)
Intolerable gastrointestional side effects (Gastrointestinal disorders) | 3 (3) | 0 (0)
injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gallstones (Gastrointestinal disorders) | 1 (1) | 0 (0)
fall (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=35) | Placebo (N=33)
protocol deviation (Investigations) | 1 (1) | 0 (0)
elective back surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Family issues (Investigations) | 1 (1) | 0 (0)
Decided to withdraw (Investigations) | 0 (0) | 6 (6)

LIMITATIONS AND CAVEATS:
Major limitation: the experimental groups were relatively small. In addition, 31% of individuals randomized to liraglutide discontinued participation. Other studies suggest tolerance of GLP-1 receptor agonists may vary by population characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No